CLINICAL TRIAL: NCT04244747
Title: The Hormonal Milieu With Different Methods of Labour Induction: a Prospective Randomized Controlled Trial
Brief Title: Labor Induction After Cesarean Section: Outcome, Hormonal Trends
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Western Galilee Hospital-Nahariya (Other Government)
Responsible Party: Principal Investigator, Dr. Maya Wolf, Head of fetal-maternal unit, Western Galilee Hospital-Nahariya
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 0190-15-NHR
Record Dates: First submitted 2019-12-19; First posted 2020-01-28 (Actual); Last update posted 2021-04-13 (Actual); Status verified 2021-04

CONDITIONS: Induction of Labor; Previous Cesarean Section; Hormonal Changes
Keywords: labor induction,; previous caesarean section; hormonal levels; breast stimulation; intracervical balloon

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- induction of labour by breast stimulation (Active Comparator): women at term with previous cesarean section and an indication to induce labor. In order to induce labour by breast stimulation, an electrical pump was used. The cup was alternated between the nipples every 15 minutes, with a pause of 15 minutes after each 30 minutes, with a total induction time of 6 hours.
  Interventions: Device: induction of labor by breast stimulation
- induction of labour by catheter balloon (Active Comparator): women at term with previous cesarean section and an indication to induce labor. In the catheter balloon group, a 16-F Foley catheter was inserted into the cervical canal and inflated with 60 cc sterile saline solution and was kept in place for 12 hours.
  Interventions: Device: induction of labor by catheter balloon
- spontaneous labour (No Intervention): women in latent phase of spontaneous labour .

INTERVENTIONS:
Device: induction of labor by breast stimulation
  Other Names: breast stimulation
  Arms: induction of labour by breast stimulation
Device: induction of labor by catheter balloon
  Other Names: catheter balloon
  Arms: induction of labour by catheter balloon

SUMMARY:
Objectives- To compare changes in labour-associated maternal and fetal hormone levels during breast stimulation, balloon induction and spontaneous labour. To compare efficacy and safety of labour induction methods in women with previous caesarean section.

Design- Participants were randomized to undergo induction of labour by breast stimulation or intracervical balloon compared to spontaneous labour (controls).

Setting- A single tertiary hospital Population- women at term, with previous caesarean section

DETAILED DESCRIPTION:
Maternal serum levels of oxytocin, prostaglandin F2α, prostaglandin E2, prolactin, estradiol and cortisol levels were analyzed at 0, 3 and 6 hours post induction initiation, including the two groups catheter balloon and breast stimulation and controls in spontaneous labor. Fetal umbilical cord hormones were measured in the three mentioned above groups. Clinical outcomes were documented in the two induction groups.

ELIGIBILITY:
Inclusion Criteria

* uncomplicated pregnancy
* 37-42 weeks of pregnancy
* singleton pregnancy
* cephalic presentation
* previous one low transverse cesarean section
* indicated induction of labour

Exclusion Criteria

* fetal anomaly
* past uterine rupture
* previous preterm cesarean section
* multiple pregnancy
* polyhydramnios
* any contraindication for vaginal delivery or catheter balloon insertion

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — women at term pregnancy
Enrollment: 100 (Estimated)
Dates: Start 2016-01 (Actual); Primary Completion 2018-07 (Actual); Study Completion 2020-01-01 (Actual)

PRIMARY OUTCOMES:
changes in labour-associated maternal and fetal hormone levels | at 0, 3 and 6 hours post induction initiation or at controls during the latent phase
  Maternal serum levels of:
  oxytocin (pg/mL)
  were analyzed at 0, 3 and 6 hours post induction initiation (T1, T2, T3) - in two induction groups: catheter balloon and breast stimulation groups the above mentioned parameter was measured also in the third study group: women in their latent phase admitted to the delivery room - the parameter was measured at 0,3,6 hours post admission this parameter was also measured in fetal umbilical cord (F) in women of the three study groups each parameter presented above were reported separately for each group (median at T1, T2, T3 and F) and compared between the three groups inter and intra groups changes were examined
changes in labour-associated maternal and fetal hormone levels | at 0, 3 and 6 hours post induction initiation or at controls during the latent phase
  Maternal serum levels of:
  prostaglandin F2α (pg/mL) were analyzed at 0, 3 and 6 hours post induction initiation (T1, T2, T3) - in two induction groups: catheter balloon and breast stimulation groups the above mentioned parameter was measured also in the third study group: women in their latent phase admitted to the delivery room - the parameter was measured at 0,3,6 hours post admission this parameter was also measured in fetal umbilical cord (F) in women of the three study groups each parameter presented above were reported separately for each group (median at T1, T2, T3 and F) and compared between the three groups inter and intra groups changes were examined
changes in labour-associated maternal and fetal hormone levels | at 0, 3 and 6 hours post induction initiation or at controls during the latent phase
  Maternal serum levels of:
  prostaglandin E2 (pg/mL) were analyzed at 0, 3 and 6 hours post induction initiation (T1, T2, T3) - in two induction groups: catheter balloon and breast stimulation groups the above mentioned parameter was measured also in the third study group: women in their latent phase admitted to the delivery room - the parameter was measured at 0,3,6 hours post admission this parameter was also measured in fetal umbilical cord (F) in women of the three study groups each parameter presented above were reported separately for each group (median at T1, T2, T3 and F) and compared between the three groups inter and intra groups changes were examined
changes in labour-associated maternal and fetal hormone levels | at 0, 3 and 6 hours post induction initiation or at controls during the latent phase
  Maternal serum levels of:
  prolactin (mclU/ml) were analyzed at 0, 3 and 6 hours post induction initiation (T1, T2, T3) - in two induction groups: catheter balloon and breast stimulation groups the above mentioned parameter was measured also in the third study group: women in their latent phase admitted to the delivery room - the parameter was measured at 0,3,6 hours post admission this parameter was also measured in fetal umbilical cord (F) in women of the three study groups each parameter presented above were reported separately for each group (median at T1, T2, T3 and F) and compared between the three groups inter and intra groups changes were examined
changes in labour-associated maternal and fetal hormone levels | at 0, 3 and 6 hours post induction initiation or at controls during the latent phase
  Maternal serum levels of:
  estradiol (pmol/L) were analyzed at 0, 3 and 6 hours post induction initiation (T1, T2, T3) - in two induction groups: catheter balloon and breast stimulation groups the above mentioned parameter was measured also in the third study group: women in their latent phase admitted to the delivery room - the parameter was measured at 0,3,6 hours post admission this parameter was also measured in fetal umbilical cord (F) in women of the three study groups each parameter presented above were reported separately for each group (median at T1, T2, T3 and F) and compared between the three groups inter and intra groups changes were examined
changes in labour-associated maternal and fetal hormone levels | at 0, 3 and 6 hours post induction initiation or at controls during the latent phase
  Maternal serum levels of:
  cortisol (μGr/dL) were analyzed at 0, 3 and 6 hours post induction initiation (T1, T2, T3) - in two induction groups: catheter balloon and breast stimulation groups the above mentioned parameter was measured also in the third study group: women in their latent phase admitted to the delivery room - the parameter was measured at 0,3,6 hours post admission this parameter was also measured in fetal umbilical cord (F) in women of the three study groups each parameter presented above were reported separately for each group (median at T1, T2, T3 and F) and compared between the three groups inter and intra groups changes were examined
changes in labour-associated maternal and fetal hormone levels | at 0, 3 and 6 hours post induction initiation or at controls during the latent phase
  Maternal serum levels of:
  testosterone (nmol/L) were analyzed at 0, 3 and 6 hours post induction initiation (T1, T2, T3) - in two induction groups: catheter balloon and breast stimulation groups the above mentioned parameter was measured also in the third study group: women in their latent phase admitted to the delivery room - the parameter was measured at 0,3,6 hours post admission this parameter was also measured in fetal umbilical cord (F) in women of the three study groups each parameter presented above were reported separately for each group (median at T1, T2, T3 and F) and compared between the three groups inter and intra groups changes were examined

SECONDARY OUTCOMES:
To compare efficacy and safety of labour induction methods in women with previous caesarean section | at birth
  the following clinical parameters were measured during the induction process or after delivery in the two induction groups (catheter balloon and breast stimulation): induction to delivery interval time in hours were measured after delivery in the two groups, medians were compared
To compare efficacy and safety of labour induction methods in women with previous caesarean section | at birth
  the following clinical parameters were measured during the induction process or after delivery in the two induction groups (catheter balloon and breast stimulation): fetal apgar score, medians were compared between the two induction groups
To compare efficacy and safety of labour induction methods in women with previous caesarean section | at birth
  the following clinical parameters were measured during the induction process or after delivery in the two induction groups (catheter balloon and breast stimulation):admission to neonatal intensive care unit rate, rates were measured after delivery and compared between the two induction groups
To compare efficacy and safety of labour induction methods in women with previous caesarean section | at birth
  the following clinical parameters were measured during the induction process or after delivery in the two induction groups (catheter balloon and breast stimulation):admission to neonatal intensive uterine rupture rates were compared in the two induction groups after delivery

CONTACTS AND LOCATIONS:
Overall Officials: Maya Wolf, MD, Principal Investigator — Galilee Medical Center, Bar-Ilan University
Locations (1):
- Galil Medical Center, Nahariya, Israel

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Kota SK, Gayatri K, Jammula S, Kota SK, Krishna SV, Meher LK, Modi KD. Endocrinology of parturition. Indian J Endocrinol Metab. 2013 Jan;17(1):50-9. doi: 10.4103/2230-8210.107841. PMID 23776853
- [Background] Mears K, McAuliffe F, Grimes H, Morrison JJ. Fetal cortisol in relation to labour, intrapartum events and mode of delivery. J Obstet Gynaecol. 2004 Feb;24(2):129-32. doi: 10.1080/01443610410001645389. PMID 14766445
- [Background] Takahata K, Horiuchi S, Tadokoro Y, Shuo T, Sawano E, Shinohara K. Effects of breast stimulation for spontaneous onset of labor on salivary oxytocin levels in low-risk pregnant women: A feasibility study. PLoS One. 2018 Feb 15;13(2):e0192757. doi: 10.1371/journal.pone.0192757. eCollection 2018. PMID 29447299
- [Background] West HM, Jozwiak M, Dodd JM. Methods of term labour induction for women with a previous caesarean section. Cochrane Database Syst Rev. 2017 Jun 9;6(6):CD009792. doi: 10.1002/14651858.CD009792.pub3. PMID 28599068
- [Background] Harper LM, Cahill AG, Boslaugh S, Odibo AO, Stamilio DM, Roehl KA, Macones GA. Association of induction of labor and uterine rupture in women attempting vaginal birth after cesarean: a survival analysis. Am J Obstet Gynecol. 2012 Jan;206(1):51.e1-5. doi: 10.1016/j.ajog.2011.09.022. Epub 2011 Sep 24. PMID 22000899
- [Background] Huisman CMA, Ten Eikelder MLG, Mast K, Oude Rengerink K, Jozwiak M, van Dunne F, Duvekot JJ, van Eyck J, Gaugler-Senden I, de Groot CJM, Franssen MTM, van Gemund N, Langenveld J, de Leeuw JW, Oude Lohuis EJ, Oudijk MA, Papatsonis D, van Pampus M, Porath M, Rombout-de Weerd S, van Roosmalen JJ, van der Salm PCM, Scheepers HCJ, Sikkema MJ, Sporken J, Stigter RH, van Wijngaarden WJ, Woiski M, Mol BWJ, Bloemenkamp KWM; PROBAAT-S project group. Balloon catheter for induction of labor in women with one previous cesarean and an unfavorable cervix. Acta Obstet Gynecol Scand. 2019 Jul;98(7):920-928. doi: 10.1111/aogs.13558. Epub 2019 Mar 7. PMID 30723900
- [Background] Singh N, Tripathi R, Mala YM, Yedla N. Breast stimulation in low-risk primigravidas at term: does it aid in spontaneous onset of labour and vaginal delivery? A pilot study. Biomed Res Int. 2014;2014:695037. doi: 10.1155/2014/695037. Epub 2014 Nov 27. PMID 25525601
- [Background] Kehl S, Weiss C, Rath W. Balloon catheters for induction of labor at term after previous cesarean section: a systematic review. Eur J Obstet Gynecol Reprod Biol. 2016 Sep;204:44-50. doi: 10.1016/j.ejogrb.2016.07.505. Epub 2016 Aug 3. PMID 27521597
- [Background] Jozwiak M, van de Lest HA, Burger NB, Dijksterhuis MG, De Leeuw JW. Cervical ripening with Foley catheter for induction of labor after cesarean section: a cohort study. Acta Obstet Gynecol Scand. 2014 Mar;93(3):296-301. doi: 10.1111/aogs.12320. Epub 2014 Jan 13. PMID 24354335
- [Background] Rahm VA, Hallgren A, Hogberg H, Hurtig I, Odlind V. Plasma oxytocin levels in women during labor with or without epidural analgesia: a prospective study. Acta Obstet Gynecol Scand. 2002 Nov;81(11):1033-9. doi: 10.1034/j.1600-0412.2002.811107.x. PMID 12421171
- [Background] Miller N, Asali AA, Agassi-Zaitler M, Neumark E, Eisenberg MM, Hadi E, Elbaz M, Pasternak Y, Fishman A, Biron-Shental T. Physiological and psychological stress responses to labor and delivery as expressed by salivary cortisol: a prospective study. Am J Obstet Gynecol. 2019 Oct;221(4):351.e1-351.e7. doi: 10.1016/j.ajog.2019.06.045. Epub 2019 Jun 27. PMID 31254523
- [Derived] Wolf MF, Sgayer I, Asslan A, Palzur E, Shnaider O, Bornstein J. The Hormonal Milieu by Different Labor Induction Methods in Women with Previous Cesarean Section: a Prospective Randomized Controlled Trial. Reprod Sci. 2021 Dec;28(12):3562-3570. doi: 10.1007/s43032-021-00667-3. Epub 2021 Jul 6. PMID 34231178